CLINICAL TRIAL: NCT01649167
Title: Longitudinal Measures of Leptin in Pregnant Women Who Developed Preeclampsia
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Researcher of the Medical Research Center (CICMED), Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: MACSSD042010
Record Dates: First submitted 2012-07-17; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: High-Risk Pregnancy
Keywords: body mass index; gestational diabetes; leptin; obesity; pregnancy.
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Overweight/obesity: Pregnant women with overweight/obesity
- gestational diabetes: Pregnant women with gestational diabetes
- normal weight: Pregnant women with normal weight

SUMMARY:
Background: Obesity in pregnancy is increasing and is a risk factor for metabolic pathology such as preeclampsia. Leptin is an adipokine which has a direct relationship to obesity.

Aim: to measure leptin in lean, obese and diabetic pregnant women at three months intervals throughout their pregnancies.

Methods: Pregnant women were recruited in the 1st trimester of pregnancy, and three groups were formed: a) with pregestational Body Mass Index (BMI) less than 25 kg/m2, b) BMI higher than 25 kg/m2 and c) with Gestational Diabetes Mellitus (GDM). Serum levels of leptin were measured with radioimmunoassay (RIA) technique.

DETAILED DESCRIPTION:
1. Introduction Obesity and type 2 diabetes (2DM) are worldwide health issues, and the incidences of both diseases are increasing rapidly. Recent research has shown that maternal nutrition during pregnancy may have long-term metabolic consequences in offspring. Many pregnant women are obese (body mass index (BMI) > 30 kg/m2). The prevalence of maternal obesity is rising, up to 20% in some antenatal clinics, which is in line with the prevalence of obesity in the general population. Obesity in pregnancy has been linked to several adverse pregnancy outcomes, including spontaneous abortion, preeclampsia, gestational diabetes (GDM), fetal macrosomia, cesarean delivery, and wound complications post-cesarean section. Both intrapartum and postpartum management of obese gravidas require multidisciplinary consultations between obstetricians, anesthesiologists, nurses, and pediatricians in order to improve the pregnancy outcomes of the mother and neonate. The American College of Obstetricians and Gynecologists (ACOG) and several authors currently support risk-reducing strategies for obese pregnant patients including limiting weight gain.

Preeclampsia is a multisystem disorder characterized by pregnancy-induced or gestational hypertension and new-onset proteinuria during the second half of pregnancy.

The aim of this study was to measure leptin in lean, obese and diabetic pregnant women at three-month intervals throughout their pregnancies to determine if this hormone could serve as a prognostic marker for preeclampsia risk.

Recruitment Women were recruited at their first visit at 10-15 weeks gestation. They were asked to attend after an overnight fast and were tested between 0700 and 0900 h. Three groups of pregnant women were formed: a) normal weight (pregestational (PG) BMI < 25 kg/m2), b) overweight-obese (PGBMI ≥ 25 kg/m2) and c) hyperglycemic in the first trimester of pregnancy confirmed as GDM in women previously known to be normoglycemic. Positive cases for preeclampsia were then subdivided.

Clinical follow-up Three examinations were performed in the 1st, 2nd, and 3rd trimesters. In each visit, the women were weighed. Blood pressure (BP) was recorded at each visit using a standard sphygmomanometer and appropriately sized cuff. If diagnosed with pregnancy-induced hypertension, the women were hospitalized and clinically supervised with an electronic monitor (Mercury, Mennem Medical) until the diagnosis of preeclampsia was confirmed or excluded.

Laboratory During each consult, blood samples were collected in Vacutainer tubes after a fasting period of 8 hours and centrifuged to separate the plasma from serum. The investigators measured albumin (mg/dl), cholesterol (mg/dl), creatinine (mg/dl), glucose (mg/dl), triglycerides (mg/dl), uric acid (mg/dl), liver enzymes (Dimension Rx L Max, Dade Behring), and hemoglobin (g/dl) (Advia 120, Bayer Health) and performed a general urine test (URiSCAN Pro). These tests were measured in the HMPMP according to standardized procedures recommended by the International Federation of Clinical Chemistry and Laboratory Medicine (IFCC).

Diagnosis of GDM At the time of recruitment, women with hyperglycemia who fulfilled the criteria and were recently diagnosed with diabetes were included in the same group as those women who were submitted to an OGT after 24 weeks' gestation and confirmed to have GDM because they had normal values of glucose prior to their pregnancies.

During pregnancy follow-up, gynecologists at the obstetric outpatient clinic used the following risk factors to screen women for GDM: a first-degree relative with diabetes, a history of GDM or macrosomia, a suspicion of macrosomia in the current pregnancy, persistent glucosuria, a rapid or excessive weight gain during early pregnancy, obesity or a random plasma glucose ≥ 7.0 mmol/l. Women with one or more of these factors underwent the standard 100 g 3-h OGTT after an overnight fast (solution provided by Laboratorio Silanes).

The diagnosis of GDM was made according to the National Diabetes Data Group (NDDG) criteria (≥ 2 abnormal values; glucose concentrations of ≥ 5.8 mmol/l for fasting, ≥ 10.6 mmol/l at 1 h, ≥ 9.2 mmol/l at 2 h, and ≥ 8.1 mmol/l at 3 h) [16].

In women with GDM, the therapeutic aims were blood glucose levels before meals < 5.0 mmol/l and 2 h postprandial < 6.5 mmol/l. If two blood glucose levels in one to two weeks were above these aims despite adequate dietary measures, then insulin of the rapid type was started or doses were increased. If these measures were insufficient to reach the therapeutic aims, then basal insulin was added.

Preeclampsia was diagnosed and classified according to the criteria specified by the technical bulletin of the ACOG and the National High Blood Pressure Education Program (NHBPEP) Working Group Report on High Blood Pressure in Pregnancy. Hypertension was described as an increase of 30 mm Hg systolic or 15 mm Hg diastolic BP as compared to the values before 20 weeks of pregnancy, or an absolute BP > 140/90 mm Hg after 20 weeks gestation if the earlier values were unknown.

Leptin Serum levels of leptin (Millipore/Linco., USA, Cat. HL-8IHK) and adiponectin (Millipore/Linco., USA, Cat. No. HADP-61HK) were determined by means of a double antibody radioimmunoassay (RIA) using materials and protocols supplied by the provider (Millipore/Linco., USA, Cat. HL-8IHK). All samples of each trimester were assayed simultaneously. The assays were run according to the manufacturer's recommendations.

Statistical analysis It was used the SPSS version 16. Continuous variables were expressed in means ± standard deviation (SD). Kruskal Wallis and Mann-Whitney U tests were considered statistically significant with a P value ≤ 0.05. Receiver Operating Characteristic (ROC) curves were used with each variable and in the cases of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Women in the first trimester of pregnancy who sought medical attention at the HMPMP, between 16 and 46 years of age with a singleton gestation.

Exclusion Criteria:

* A previously known chronic metabolic disease (diabetes, pregestational dyslipidemia, hypertension, collagen vascular diseases, inflammatory bowel disease and chronic inflammatory conditions, or corticosteroid use).

Ages: 16 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who had received medical attention during pregnancy at the HMPMP in Toluca, Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-02; Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verónica Jackeline García Solorio, MSc, Principal Investigator — Autonomous University of the State of Mexico; Hugo Mendieta Zerón, PhD, Study Chair — Autonomous University of the State of Mexico